CLINICAL TRIAL: NCT02025634
Title: Determining the Efficacy of Intravenous Acetaminophen as a Non-Narcotic Postoperative Pain Management Technique Following Knee Arthroscopy
Brief Title: Intravenous Acetaminophen for Non-Narcotic Postoperative Pain Management Following Knee Arthroscopy
Acronym: IVTYLENOL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: University of Central Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 503526
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Pain, Postoperative
Keywords: Pain, Postoperative; Ofirmev; Acetaminophen; Analgesics, Non-Narcotic; Arthroscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous acetaminophen (Experimental): Infusion of Intravenous acetaminophen (Ofirmev)
  Interventions: Drug: Intravenous Acetaminophen
- Placebo (0.9% Normal Saline Infusion) (Placebo Comparator): Infusion of 100 ml of 0.9 NS Normal Saline
  Interventions: Drug: Placebo (0.9% Normal Saline infusion)

INTERVENTIONS:
Drug: Intravenous Acetaminophen — Participants randomized to intravenous acetaminophen (Ofirmev) will receive an infusion of Ofirmev in 100 ml of 0.9 NS according to manufacturer's recommendations related to subject's weight.
  Other Names: Ofirmev
  Arms: Intravenous acetaminophen
Drug: Placebo (0.9% Normal Saline infusion) — Infusion of 100 ml of 0.9% NS
  Other Names: NS
  Arms: Placebo (0.9% Normal Saline Infusion)

SUMMARY:
The purpose of this randomized, placebo controlled, single blind study is to determine if postoperative pain levels, as measured by a verbal numeric pain rating scale (VNRS), are reduced with the administration of IV acetaminophen when compared to a control group. Particular focus will be on the postoperative opioid consumption. In addition, we will ascertain if the total time the participant is in the PACU differs in those who receive the IV acetaminophen versus those who do not.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled, single blind study of intravenous (IV) acetaminophen in a postoperative arthroscopy patient population. Although use of this medication as a non-narcotic analgesia has been validated in other patient populations such as post operative pelvic and abdominal surgeries, it has not been demonstrated in those who have recently undergone knee arthroscopy with or without chondroplasty. In this study all participants will be injected with a standard of care intra-articular dose of ropivacaine HCl, .2% (Naropin) prior to transfer to the Post Anesthesia Care Unit (PACU). Each will be randomized 1:1 to receive IV acetaminophen in 100ml of 0.9% NS (treatment group) or a 100 ml 0.9 % NS placebo (control).

The PACU nursing staff will periodically ascertain the participants' pain scores on a 0-10 scale. All other pain medication or related treatment will be recorded. Statistical analysis will be done to determine if there is a difference in pain scores between the treatment versus control group. Further evaluation will examine if opioid consumption and total time in PACU differs between groups.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled for knee arthroscopy with or without chondroplasty.
* Scheduled arthroscopy procedure will not include ligament repairs or ligament reconstructions and/or bone cutting or fixation procedures.
* Has not received any acetaminophen (IV, PR, PO) within at least 8 hours of the initiation of surgery.
* Is willing and able to sign an informed consent.

Exclusion Criteria:

* Is undergoing arthroscopy for ligament repairs/reconstructions and bone cutting or fixation procedures
* Has self-reported and/or documented previous hypersensitivity to acetaminophen.
* Has self-reported and/or documented history of hepatic disease or impairment.
* Pre-operative calculated creatinine clearance (CrCL) less than 40 ml/min.
* Has a medical history of alcohol abuse and/or currently drinks more than 3 alcoholic beverages per day.
* Has a medical history of substance dependence (i.e. prescription analgesics or illegal drugs such as cocaine, heroin, etc…). May be self-reported or maybe per the judgment of the physician PI/Sub-I.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2013-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Homan, DO, Principal Investigator — Florida Hospital Celebration Health
Locations (1):
- Florida Hospital Celebration Health, Celebration, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion)
Started | 65 | 54
Completed | 65 | 54
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion) | Total
Number analyzed (Participants) | 65 | 54 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 34 | 74
  >=65 years | 25 | 20 | 45
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 66
  Male | 31 | 22 | 53
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Levels
Description: To determine if postoperative pain levels, as measured by a Verbal Numerical Rating Scale (VNRS), are reduced with the administration of IV acetaminophen when compared to a control group. In the VNRS, the user has the option to verbally rate their scale from 0 to 10. Zero indicates the absence of pain, while 10 represents the most intense pain possible.
Time Frame: up to 8 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion)
Number analyzed (Participants) | 65 | 54
score on a scale | 1.3160 (1.33510) | 2.1362 (1.59323)

2. Secondary Outcome: Postoperative Opioid Consumption
Description: To learn if opioid consumption is reduced when IV acetaminophen is provided immediately post-operatively.
Time Frame: up to 8 hours
Measure: Mean (Full Range); unit: mg
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion)
Number analyzed (Participants) | 65 | 54
mg | 3 [0 to 50] | 2 [0 to 28.1]

3. Other Pre Specified Outcome: Total Time in Post Anesthesia Care Unit (PACU) (or "Recovery Room")
Description: To ascertain if the total time the participant remains in the PACU (from admission to discharge) differs between those who received IV acetaminophen versus those who do not receive IV acetaminophen.
Time Frame: up to 8.6 hours
Measure: Mean (Full Range); unit: hours
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion)
Number analyzed (Participants) | 65 | 54
hours | 3.30 [1.08 to 5.22] | 3.40 [1.23 to 8.60]

ADVERSE EVENTS:
Arm/Group | Intravenous Acetaminophen | Placebo (0.9% Normal Saline Infusion)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/54
Other Adverse Events (participants affected / at risk) | 0/65 | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes